CLINICAL TRIAL: NCT04196491
Title: A Phase 1, Open-label, Multicenter Study to Evaluate the Safety of bb2121 in Subjects With High Risk, Newly Diagnosed Multiple Myeloma (KarMMa-4)
Brief Title: A Study to Evaluate the Safety of bb2121 in Subjects With High Risk, Newly Diagnosed Multiple Myeloma (NDMM)
Acronym: KarMMa-4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BB2121-MM-004; U1111-1243-5088 (Other: WHO)
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Newly diagnosed multiple myeloma; BB2121; KarMMa-4; Phase I; NDMM; High Risk; R-ISS III; KRd; RVd; Dara-KRd; Dara-RVd; CyBorD; BCMA
MeSH Terms: conditions — Multiple Myeloma | interventions — idecabtagene vicleucel; fludarabine; Cyclophosphamide; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): * bb2121 autologous CAR T cells will be infused at a dose ranging from 150 - 800 x 10^6 CAR+ T cells after receiving lymphodepleting chemotherapy with a planned starting dose of 450 x 10^6 CAR+ T cells.
  * Lenalidomide maintenance therapy is recommended for all patients and should be initiated upon adequate bone marrow recovery or from 90-day post-bb2121 infusion, whichever is later
  Interventions: Biological: bb2121; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Lenalidomide

INTERVENTIONS:
Biological: bb2121 — CAR-T Cell Therapy
  Other Names: ide-cel
Drug: Fludarabine — Lymphodepleting Chemotherapy
Drug: Cyclophosphamide — Lymphodepleting Chemotherapy
Drug: Lenalidomide — Maintenance Therapy

SUMMARY:
This is a multicenter, open-label, phase 1, single arm study intended to determine the optimal target dose and safety of bb2121 in subjects with HR (R-ISS Stage III per IMWG criteria) NDMM. Subjects should have received 3 Cycles of standard induction therapy prior to undergoing leukapheresis procedure to collect autologous mononuclear cells for manufacture of the drug product (bb2121). Following manufacture of the drug product, subjects will receive fourth cycle of induction therapy followed by lymphodepleting therapy with fludarabine and cyclophosphamide prior to bb2121 infusion. Maintenance therapy is recommended for all subjects who have received bb2121 infusion and should be initiated upon adequate bone marrow recovery or from 90-day post-bb2121 infusion, whichever is later.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy all of the following criteria to be enrolled in the study:

1. Subject is newly diagnosed and has symptomatic Multiple Myeloma (MM) prior to initiating induction anti-myeloma therapy
2. Subject is ≥ 18 years of age at the time of initial diagnosis of MM
3. Subject has measurable disease at initial diagnosis by

   * M-protein and/or
   * Light chain MM without measurable disease in the serum or urine
4. Subject has high-risk MM at the time of initial diagnosis of MM per R-ISS Stage III as defined by IMWG:

   * ISS Stage III and cytogenetic abnormalities with t(4; 14) and/or del(17p); and/or t(14:16) by iFISH; or;
   * ISS Stage III and serum LDH > ULN
5. Subject has Eastern Cooperative Oncology Group performance ≤ 1
6. Subjects has received ≤ to 3 cycles of the following induction anti-myeloma therapy prior to enrollment:

   * Cycle 1: one of the following regimens (RVd, KRd, CyBorD, D-RVd and D-KRd)
   * Cycle 2 to Cycle 3: either KRd or RVd (Cycle 3 must be without dexamethasone)

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment: The presence of any of the following will exclude a subject from enrollment:

At initial diagnosis, screening and prior to initiation of induction therapy for MM:

1. Subject has non-secretory MM

   During Screening:
2. Subject received any treatments for MM other than up to 3 cycles of induction therapy per protocol
3. Subject has any of the following laboratory abnormalities:

   1. Absolute neutrophil count < 1,000/μL
   2. Platelet count < 50,000 mm3
   3. Hemoglobin < 8 g/dL (< 4.9 mmol/L)
   4. Serum creatinine clearance < 45 mL/min
   5. Corrected serum calcium > 13.5 mg/dL (> 3.4 mmol/L)
   6. Serum aspartate aminotransferase or alanine aminotransferase > 2.5 × upper limit of normal
   7. Serum total bilirubin > 1.5 × ULN or > 3.0 mg/dL for subjects with documented Gilbert's syndrome
   8. INR or aPTT > 1.5 × ULN
4. Subject has history or presence of clinically significant CNS pathology
5. Subjects has high risk for developing deep vein thrombosis or pulmonary embolus and are unable or unwilling to undergo anti-thrombotic therapy
6. Subject has peripheral neuropathy of > Grade 2 severity according to the NCI CTCAE Version 4.03 with bortezomib based induction regimen
7. Subjects has moderate or severe pulmonary hypertension
8. Subject has intolerance to components of induction regimen (KRd or RVd) or has any contraindication to one or the other drug
9. Subject has not recovered from induction therapy-related toxicities (non-hematologic) to < grade 1 CTCAE at the time of screening
10. Subject has prior history of deep vein thrombosis or pulmonary embolus (PE) within 6 months of starting study treatment
11. Subject has cardiac conditions such as:

    1. Echocardiogram or multi gated acquisition assessment of left ventricular ejection fraction < 45%
    2. Subject has a history of clinically significant cardiovascular disease or clinically significant ECG abnormalities
12. Subject has Pulmonary conditions such as:

    1. Subject has known chronic obstructive pulmonary with a forced expiratory vol in 1 sec 50% of predicted normal.
    2. Inadequate pulmonary function defined as oxygen saturation < 92 % on room air
13. Subject needs ongoing treatment with chronic immunosuppressants
14. Subject has history of primary immunodeficiency
15. Subject is seropositive for human immunodeficiency virus, chronic or active hepatitis B or active hepatitis A or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) rates | Up to completion of DLT period after last subject bb2121 infused
  DLTs will be assessed during the DLT interval (ie, within 21 days immediately after bb2121 infusion). DLTs are defined as any bb2121 related Grade 3 to 5 toxicity.
Adverse Events (AEs) | Approximately 2 years after last subject bb2121 infused
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE.

SECONDARY OUTCOMES:
Proportion of subjects who achieved Complete Response (CR) Rate | Approximately 2 years after last subject bb2121 infused
  Is defined as proportion of subjects who achieved CR or better according to IMWG Uniform Response Criteria for Multiple Myeloma for multiple myeloma will be determined by an Investigator assessment.
Overall Response Rate (ORR) | Approximately 2 years after last subject bb2121 infused
  Is defined as proportion of subjects who achieved PR or better according to IMWG Uniform Response Criteria for Multiple Myeloma as determined by an Investigator assessment
Duration of Response (DoR) | Approximately 2 years after last subject bb2121 infused
  Is defined as time from first documentation of response (PR or better) to first documentation of progressive disease (PD) or death from any cause, whichever occurs first, for responders.
Time to Complete Response (TCR) | Approximately 2 years after last subject bb2121 infused
  Is defined as time from bb2121 infusion date to first documentation of CR for responders (Complete Response (CR) or better).
Time to start maintenance | Approximately 2 years after last subject bb2121 infused
  Is defined as time to start lenalidomide maintenance therapy post-bb2121 infusion
Feasibility of initiating maintenance | Approximately 2 years after last subject bb2121 infused
  Number of subjects starting the maintenance or on maintenance between D90 and D110
Progression-free Survival (PFS) | Approximately 2 years after last subject bb2121 infused
  Is defined as time from bb2121 infusion date to first documentation of PD, or death due to any cause, whichever occurs first.
Overall Survival (OS) | Approximately 2 years after last subject bb2121 infused
  Is defined as time from bb2121 infusion date to time of death due to any cause
Pharmacokinetics - Cmax | Approximately 2 years after last subject bb2121 infused
  Maximum transgene level
Pharmacokinetics - Tmax | Approximately 2 years after last subject bb2121 infused
  Time to peak transgene level
Pharmacokinetics - AUC | Approximately 2 years after last subject bb2121 infused
  Area under the curve of the transgene level

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (22):
- United States (22):
  - Local Institution - 119, Phoenix, Arizona
  - Local Institution - 110, Los Angeles, California
  - Local Institution - 116, San Francisco, California
  - Local Institution - 106, Denver, Colorado
  - Local Institution - 101, Jacksonville, Florida
  - Local Institution - 113, Tampa, Florida
  - Local Institution - 108, Atlanta, Georgia
  - Local Institution - 123, Atlanta, Georgia
  - Local Institution - 115, Boston, Massachusetts
  - Local Institution - 122, Boston, Massachusetts
  - Local Institution - 117, Hackensack, New Jersey
  - Local Institution - 121, New York, New York
  - Local Institution - 109, New York, New York
  - Local Institution - 124, New York, New York
  - Local Institution - 120, Charlotte, North Carolina
  - Local Institution - 112, Portland, Oregon
  - Local Institution - 118, Philadelphia, Pennsylvania
  - Local Institution - 103, Nashville, Tennessee
  - Local Institution - 102, Dallas, Texas
  - Local Institution - 114, Houston, Texas
  - Local Institution - 104, Seattle, Washington
  - Local Institution - 107, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- [Derived] Parmar H, Vesole DH, Biran N. From VAD to VRD: Is Transplant Still Needed in the Upfront Setting of Myeloma? Cancer J. 2021 May-Jun 01;27(3):190-195. doi: 10.1097/PPO.0000000000000522. PMID 34549906
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome